CLINICAL TRIAL: NCT01489826
Title: A Phase 1, Pharmacokinetically-Guided, Dose Escalation Study to Assess the Safety and Tolerability of Dexanabinol in Patients With Advanced Solid Tumours
Brief Title: A Phase 1 Study of Dexanabinol in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: e-Therapeutics PLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETS2101-001
Record Dates: First submitted 2011-12-07; First posted 2011-12-12 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-10

CONDITIONS: Solid Tumour
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — HU 211; cremophor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Dexanabinol 2 mg/kg (Experimental): Dexanabinol 2 mg/kg formulated in cremophor/ethanol, administered once weekly intravenously (i.v.)
  Interventions: Drug: Dexanabinol; Other: Cremophor
- Dexanabinol 3 mg/kg (Experimental): Dexanabinol 3 mg/kg formulated in cremophor/ethanol, administered once weekly intravenously (i.v.)
  Interventions: Drug: Dexanabinol; Other: Cremophor
- Dexanabinol 6 mg/kg (Experimental): Dexanabinol 6 mg/kg formulated in cremophor/ethanol, administered once weekly intravenously (i.v.)
  Interventions: Drug: Dexanabinol; Other: Cremophor
- Dexanabinol 12 mg/kg (Experimental): Dexanabinol 12 mg/kg formulated in cremophor/ethanol, administered once weekly intravenously (i.v.)
  Interventions: Drug: Dexanabinol; Other: Cremophor
- Dexanabinol 15 mg/kg (Experimental): Dexanabinol 15 mg/kg formulated in cremophor/ethanol, administered once weekly intravenously (i.v.)
  Interventions: Drug: Dexanabinol; Other: Cremophor
- Dexanabinol 22 mg/kg (Experimental): Dexanabinol 22 mg/kg formulated in cremophor/ethanol, administered once weekly intravenously (i.v.)
  Interventions: Drug: Dexanabinol; Other: Cremophor
- Dexanabinol 30 mg/kg (Experimental): Dexanabinol 30 mg/kg formulated in cremophor/ethanol, administered once weekly intravenously (i.v.)
  Interventions: Drug: Dexanabinol; Other: Cremophor
- Dexanabinol 36 mg/kg (Experimental): Dexanabinol 36 mg/kg formulated in cremophor/ethanol, administered once weekly intravenously (i.v.)
  Interventions: Drug: Dexanabinol; Other: Cremophor
- Dexanabinol Expansion Phase (Experimental): Dexanabinol 30 mg/kg formulated in cremophor/ethanol, administered once weekly intravenously (i.v.)
  Interventions: Drug: Dexanabinol; Other: Cremophor

INTERVENTIONS:
Drug: Dexanabinol — Patients will (initially) be given a slow intravenous (i.v.) infusion of Dexanabinol over 3 hours on Days 1, 8 and 15 of a three weekly (21 day) cycle.
  Other Names: ETS2101; HU-211
Other: Cremophor — Drug vehicle.

SUMMARY:
This study is a trial of Dexanabinol in patients with advanced solid tumours. The purposes of this protocol are to study different doses of the study drug to determine the maximum safe dose and to further understand the safety of the study drug; to understand what the body does to the study drug; to understand what the study drug does to the body and to measure any reduction in size of patients' cancer tumour(s).

Dexanabinol is a synthetic cannabinoid derivative with reduced psychotropic potential which was initially investigated as a neuroprotective agent. Because of its method of action however it is thought that it may have the effect of destroying cancer cells by reducing the level of control on networks that prevent cancer cells dying.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients defined by age ≥18 years.
2. Patients with histologically or cytologically confirmed solid tumours that are advanced, metastatic and or progressive, for whom there is no effective standard therapy available.
3. Eastern Collaborative Oncology Group (ECOG) Performance Status of ≤2.
4. Any acute or chronic adverse effects of prior chemotherapy or radiotherapy have resolved to < Grade 2 as determined by Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria, with the exception of alopecia.
5. Evaluable disease, either measurable on imaging, or with informative tumour marker(s), as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 (Eisenhauer, et al. 2009).
6. Laboratory values at Screening:

   * Absolute neutrophil count ≥1.5 x 109/L;
   * Platelets ≥100 x 109/L;
   * Total bilirubin <1.5 times the upper limit of normal;
   * Aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal;
   * Alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal;
   * Estimated glomerular filtration rate (GFR) of >50 mL/min (based on the Wright formula (Wright, et al. 2001); and
   * Negative human chorionic gonadotropin (hCG) test in women of childbearing potential (defined as women ≤50 years of age or history of amenorrhea for ≤12 months prior to study entry). Sexually active male and female patients of childbearing potential must agree to use an effective method of birth control (e.g. barrier methods with spermicides, oral or parenteral contraceptives and/or intrauterine devices) during the entire duration of the study and for 1 month after final administration of Dexanabinol, or the patient must be surgically sterile (with documentation in the patient's medical records).
7. If there is a history of treated brain metastases, these must have been clinically stable for ≥4 weeks prior to enrollment.
8. Have a life expectancy of >3 months.
9. Ability to give written, informed consent prior to any study-specific Screening procedures, with the understanding that the consent may be withdrawn by the patient at any time without prejudice.
10. Be willing and able to comply with the study protocol procedures.

Exclusion Criteria:

1. Patient is pregnant or breast feeding.
2. History of clinically significant cardiac condition, including ischemic cardiac event, myocardial infarction or unstable cardiac disease within 3 months of Cycle 1, Day 1.
3. Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to Cycle 1, Day 1. Localised palliative radiotherapy is permitted for symptom control.
4. Major surgery within 6 weeks prior to Cycle 1, Day 1.
5. Known human immunodeficiency virus positivity.
6. Active hepatitis B or C or other active liver disease (other than malignancy).
7. Use of any investigational agents within 4 weeks of Cycle 1, Day 1.
8. Any active, clinically significant, viral, bacterial, or systemic fungal infection within 4 weeks prior to Cycle 1, Day 1.
9. History of significant chronic or recurrent infections requiring treatment or any uncontrolled intercurrent illness that would jeopardize patient safety, interfere with the objectives of the protocol, or limit patient compliance with study requirements, as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Plummer, MD, Principal Investigator — Northern Centre for Cancer Care, Freeman Hospital, Newcastle-upon-Tyne, UK; Alan Anthoney, MD, Principal Investigator — Leeds Cancer Centre at St. James's University Hospital; Jeff Evans, MD, Principal Investigator — The Beatson West of Scotland Cancer Centre, 1053 Great Western Road, Glasgow
Locations (3):
- United Kingdom (3):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Northern Centre for Cancer Care, Freeman Hospital, Newcastle-upon-Tyne, UK, Newcastle upon Tyne, Tyne and Wear
  - The Beatson West of Scotland Cancer Centre,, Glasgow

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 6 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 15 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg | Dexanabinol Expansion Phase
Started | 3 | 3 | 3 | 7 | 3 | 3 | 9 | 3 | 6
Completed | 3 | 3 | 3 | 7 | 3 | 3 | 9 | 3 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dexanabinol Dose Escalation - Cohort 1; Dexanabinol Dose Escalation - Cohort 2; Dexanabinol Dose Escalation - Cohort 3; Dexanabinol Dose Escalation - Cohort 4; Dexanabinol Dose Escalation - Cohort 5; Dexanabinol Dose Escalation - Cohort 6; Dexanabinol Dose Escalation - Cohort 7; Dexanabinol Dose Escalation - Cohort 8: Open label, dose escalation phase to assess tolerability and pharmacokinetics of dexanabinol in patients with advanced tumours
- Dexanabinol Expansion Phase: Open label, expansion phase to assess pharmacodynamics of dexanabinol in patients with advanced tumours at the MTD/MAD (30 mg/kg)
- Total: Total of all reporting groups
Arm/Group | Dexanabinol Dose Escalation - Cohort 1 | Dexanabinol Dose Escalation - Cohort 2 | Dexanabinol Dose Escalation - Cohort 3 | Dexanabinol Dose Escalation - Cohort 4 | Dexanabinol Dose Escalation - Cohort 5 | Dexanabinol Dose Escalation - Cohort 6 | Dexanabinol Dose Escalation - Cohort 7 | Dexanabinol Dose Escalation - Cohort 8 | Dexanabinol Expansion Phase | Total
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 3 | 3 | 9 | 3 | 6 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 3 | 7 | 3 | 3 | 9 | 3 | 6 | 38
  >=65 years | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (10.21) | 61.3 (7.64) | 69.0 (11.14) | 57.9 (7.27) | 52.3 (5.51) | 62.0 (13.11) | 64.6 (6.91) | 63.7 (12.70) | 56.3 (12.75) | 61.2 (9.69)
Gender [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 4 | 12
  Male | 2 | 2 | 3 | 5 | 2 | 2 | 9 | 1 | 2 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Dose Limiting Toxicity (DLT)
Description: Patients will be sequentially assigned to increasing doses of Dexanabinol, to establish the maximum tolerated dose (MTD) (highest dose it is safe to give patients) or alternatively the maximum administered dose (MAD).
  3 patients will be enrolled to a cohort to assess each dose level. Dose escalation to a cohort of 3 new patients will occur when all patients in the previous cohort have completed the first cycle i.e. the first 3 doses followed by observation through to Day 22, and no DLT has occurred. Upon occurrence of the first DLT within a cohort, an additional 3 patients were to be added to that cohort. For a six patient cohort, all 6 patients were to have completed their first dexanabinol treatment cycle with no more than 1 DLT before dose escalation to the next cohort. If 2 or more DLTs occur in a cohort, the next lower dose level will be declared the MTD.
  DLTs will be graded for severity based on the National Cancer Institute (NCI) Common Terminology Criteria version 4.03.
Time Frame: Each patient will be followed for 22 days
Population: Patients will be sequentially assigned to increasing doses of Dexanabinol, to establish the MTD (highest dose it is safe to give patients) or alternatively the Maximum Administered Dose(MAD). DLT evaluation in 3 to 6 patients at end of 1 treatment cycle
Measure: Number; unit: Number of patients with DLT
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 6 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 15 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg | Dexanabinol Expansion Phase
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 3 | 3 | 9 | 3 | 6
Number of patients with DLT | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0

2. Secondary Outcome: Area Under Curve (AUC) of Dexanabinol on Cycle 1 Day 1
Description: Geometric mean AUC of Dexanabinol (0-infinity) on Cycle 1 Day 1.
Time Frame: Cycle 1- Day 1: pre-dose (0h); 1, 2, 3 h post start of infusion; 5, 10, 15, 30 min post-end infusion; 1, 2, 3, 4, 6, 8, 10 and 24 h post-end infusion.
Population: Concentrations of dexanabinol were not reported for some patients on Days 1 or 8 (including all patients in the 6 mg/kg arm) because the bioanalytical assay, in these instances, was not appropriately validated on the day of the assay. For the purposes of the PK analysis, the results from the expansion phase arm were combined with the 30 mg/kg arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 15 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg
Number analyzed (Participants) | 2 | 1 | 4 | 2 | 3 | 7 | 1
ng.h/mL | 2620 (33.9) | 6520 (0) | 25000 (53.3) | 27500 (5.99) | 46900 (41.9) | 110000 (59.9) | 219000 (0)

3. Secondary Outcome: Maximum Concentration (Cmax) of Dexanabinol Cycle 1 Day 1
Description: Mean Cmax of Dexanabinol on Cycle 1 Day 1
Time Frame: Cycle1 - Day 1: pre-dose (0h); 1, 2, 3 h post start of infusion; 5, 10, 15, 30 min post-end infusion; 1, 2, 3, 4, 6, 8, 10 and 24 h post-end infusion.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 15 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 3 | 7 | 1
ng/mL | 606 (20.9) | 1580 (0.895) | 6950 (76.8) | 7790 (24.8) | 13000 (27.4) | 28800 (62.3) | 45600 (0)

4. Secondary Outcome: Number of Adverse Events (AEs)
Description: AEs will be graded according to the NCI CTCAE v4.03 for cancer clinical trials
Time Frame: 30 +/-3 days from the end of the last infusion
Population: The numbers represent the total number of AEs per group. Refer to AE tables for specific information.
Measure: Number; unit: Events
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 6 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 15 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg | Dexanabinol Expansion Phase
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 3 | 3 | 9 | 3 | 6
Events | 68 | 31 | 26 | 90 | 64 | 60 | 85 | 47 | 62

5. Secondary Outcome: Progression Free Survival
Description: Tumour response evaluation using RECIST 1.1. (Assessment by CT scan or MRI).
Time Frame: At Screening and after every 2 cycles of treatment (+/-1 week)
Population: Patients included in this analysis were from the 'Efficacy population', defined as those with a baseline and at least one post-baseline assessment of efficacy.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 6 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 15 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg | Dexanabinol Expansion Phase
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 6 | 2 | 6
Days | 133.0 [100.0 to 267.0] | 70.0 [36.0 to NA] — Upper inter-quartile range could not be calculated due to censored value. | 37.0 [35.0 to NA] — Upper inter-quartile range could not be calculated due to censored value. | 43.0 [36.0 to 51.0] | 176.0 [86.0 to 176.0] | 293.0 [293.0 to 293.0] | 40.5 [36.0 to 66.0] | NA [43.0 to NA] — Median could not be calculated as there were only two values. Upper inter-quartile range could not be calculated due to censored value. | 37.0 [36.0 to 49.0]

6. Secondary Outcome: Area Under Curve (AUC) of Dexanabinol on Cycle 1 Day 8
Description: Geometric mean AUC of Dexanabinol (0-infinity) on Cycle 1 Day 8.
Time Frame: Cycle 1- Day 8: pre-dose (0h); 1, 2, 3 h post start of infusion; 5, 10, 15, 30 min post-end infusion; 1, 2, 3, 4, 6, 8, 10 and 24 h post-end infusion.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg
Number analyzed (Participants) | 2 | 2 | 5 | 3 | 7 | 1
ng.h/mL | 2600 (31.5) | 5140 (2.39) | 29500 (47.2) | 45700 (40.4) | 96500 (67.2) | 145000 (0)

7. Secondary Outcome: Area Under Curve (AUC) of Cremophor on Cycle 1 Day 1
Description: Geometric mean AUC of Cremophor (0-27hour) on Cycle 1 Day 1.
Time Frame: as for outcome 2
Population: This analysis was performed on all patients who received study drug and for whom PK samples were obtained (the PK analysis population). For the purposes of the PK analysis, the results from the expansion phase arm were combined with the 30 mg/kg arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µL.h/mL
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 6 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 15 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 14 | 3
µL.h/mL | NA (NA) — Geometric mean could not be calculated, as too many values were below the level of quantification. | NA (NA) — Geometric mean could not be calculated, as too many values were below the level of quantification. | 10.3 (101) | 46.2 (69.9) | 29.5 (64.0) | 92.4 (40.5) | 120 (39.1) | 152 (75.8)

8. Secondary Outcome: Area Under Curve (AUC) of Cremophor on Cycle 1 Day 8
Description: Geometric mean AUC of Cremophor (0-27hour) on Cycle 1 Day 8.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µL.h/mL
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 6 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 15 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3 | 14 | 1
µL.h/mL | NA (NA) — Geometric mean could not be calculated, as too many values were below the level of quantification. | 3.15 (287) | 14.8 (50.1) | 43.6 (40.0) | 29.8 (88.3) | 97.1 (37.0) | 146 (54.9) | 138 (0)

9. Secondary Outcome: Maximum Concentration (Cmax) of Dexanabinol Cycle 1 Day 8
Description: Mean Cmax of Dexanabinol on Cycle 1 Day 8
Time Frame: Cycle1 - Day 8: pre-dose (0h); 1, 2, 3 h post start of infusion; 5, 10, 15, 30 min post-end infusion; 1, 2, 3, 4, 6, 8, 10 and 24 h post-end infusion.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 15 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg
Number analyzed (Participants) | 2 | 2 | 5 | 3 | 3 | 7 | 1
ng/mL | 705 (2.01) | 1410 (12.6) | 8600 (58.3) | 9560 (49.6) | 14600 (44.0) | 27800 (56.7) | 34900 (0)

10. Secondary Outcome: Maximum Concentration (Cmax) of Cremophor Cycle 1 Day 1
Description: Mean Cmax of Cremophor on Cycle 1 Day 1
Time Frame: as for outcome 3
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µL/mL
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 6 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 15 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 14 | 3
µL/mL | NA (NA) — Geometric mean could not be calculated, as too many values were below the level of quantification. | NA (NA) — Geometric mean could not be calculated, as too many values were below the level of quantification. | 1.30 (21.2) | 3.42 (46.9) | 2.72 (11.0) | 7.78 (33.3) | 8.49 (33.3) | 11.8 (37.5)

11. Secondary Outcome: Maximum Concentration (Cmax) of Cremophor Cycle 1 Day 8
Description: Mean Cmax of Cremophor on Cycle 1 Day 8
Time Frame: as for outcome 9
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µL/mL
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 6 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 15 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3 | 14 | 1
µL/mL | NA (NA) — Geometric mean could not be calculated, as too many values were below the level of quantification. | 0.754 (44.7) | 1.69 (168) | 2.99 (34.4) | 2.22 (34.2) | 8.15 (6.51) | 9.91 (31.3) | 10.1 (0)

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the day of the first dose of study drug (cycle 1 day 1) through to the final study visit (30 days +/- 3 days) after discontinuation of study drug.
Arm/Group | Dexanabinol 2 mg/kg | Dexanabinol 3 mg/kg | Dexanabinol 6 mg/kg | Dexanabinol 12 mg/kg | Dexanabinol 15 mg/kg | Dexanabinol 22 mg/kg | Dexanabinol 30 mg/kg | Dexanabinol 36 mg/kg | Dexanabinol Expansion Phase
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 1/3 | 2/7 | 2/3 | 1/3 | 5/9 | 1/3 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 7/7 | 3/3 | 3/3 | 9/9 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexanabinol 2 mg/kg (N=3) | Dexanabinol 3 mg/kg (N=3) | Dexanabinol 6 mg/kg (N=3) | Dexanabinol 12 mg/kg (N=7) | Dexanabinol 15 mg/kg (N=3) | Dexanabinol 22 mg/kg (N=3) | Dexanabinol 30 mg/kg (N=9) | Dexanabinol 36 mg/kg (N=3) | Dexanabinol Expansion Phase (N=6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Renal inpairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered state of conciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexanabinol 2 mg/kg (N=3) | Dexanabinol 3 mg/kg (N=3) | Dexanabinol 6 mg/kg (N=3) | Dexanabinol 12 mg/kg (N=7) | Dexanabinol 15 mg/kg (N=3) | Dexanabinol 22 mg/kg (N=3) | Dexanabinol 30 mg/kg (N=9) | Dexanabinol 36 mg/kg (N=3) | Dexanabinol Expansion Phase (N=6)
Nausea (Gastrointestinal disorders) | 1 (4) | 2 (2) | 0 (0) | 2 (3) | 2 (12) | 1 (1) | 2 (7) | 3 (5) | 1 (1)
Fatigue (General disorders) | 1 (3) | 0 (0) | 2 (2) | 4 (9) | 1 (3) | 0 (0) | 2 (3) | 2 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 1 (1) | 3 (10) | 1 (3) | 2 (4)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (3) | 0 (0) | 2 (2) | 2 (5) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (10) | 0 (0) | 1 (1) | 1 (1) | 2 (8) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (12) | 2 (5) | 2 (10)
Oedema peripheral (General disorders) | 2 (4) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (12) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
AST increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (12) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (7) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor (or is agents) that restricts the PIs rights to discuss or publish trial results after the trial is completed.